CLINICAL TRIAL: NCT00497432
Title: Hyperbaric Oxygen Treatment In Patients With White Matter Hyperintensities On Magnetic Resonance Imaging and Neurologic Deficits
Brief Title: Hyperbaric Oxygen Treatment in Patients With White Matter Hyperintensities
Status: Completed | Type: Observational
Sponsor: St. Luke's Hospital, Chesterfield, Missouri (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, John Davidson, Principal Investigator, St. Luke's Hospital, Chesterfield, Missouri
Other Study IDs: 2006.028
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Neurological Impairments; Leukoencephalopathies
Keywords: Hyperbaric Oxygen
MeSH Terms: conditions — Leukoencephalopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this study is to assess whether hyperbaric oxygen treatment improves neurological function in patients who exhibit white matter hyperintensities on MRI examination.

The secondary goal of this study is to determine if it is possible using MRI to discern a difference in perfusion of central nervous system tissue in regions of white matter hyperintensities after hyperbaric oxygen administration as compared to hyperbaric air.

DETAILED DESCRIPTION:
Consecutively enrolled patients will be assigned to hyperbaric oxygen or hyperbaric air by random number. Physicians supervising the hyperbaric treatments and the treating technicians, the evaluating neurologist, and the interpreter of the MRIs will be blinded regarding patient treatment status. All patients who receive placebo will be offered treatment with hyperbaric oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years of age
* White Matter Hyperintensities on MRI of brain
* Two or more symptoms and/or Neurological impairments e.g. gait disturbance, dysequilibrium, decline in cognitive function, upper motor neuron deficit, dysmetria, hyper-reflex or unilateral increase in muscle tone

Exclusion Criteria:

* Contraindications to hyperbaric oxygen therapy e.g. pulmonary emphysema or bullae, claustrophobia, seizure disorder
* Inability of the patient to tolerate pressurization e.g. eustachian tube dysfunction
* Extreme cognitive impairment
* Major Depression
* Other uncontrolled co-morbidities e.g. diabetes, hypertension, thyroid disorders, carotid artery stenosis (over 70%), renal or hepatic dysfunction
* History of brain tumor, head trauma, electroshock therapy,brain irradiation or migraine headaches

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neurological Symptom or deficits who demonstrate evidence of small vessel disease of the brain by leukoencephalopathy
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The rating scores on the physical/neurological examinations are qualitative, comparisons between the treated and the placebo groups must be analyzed utilizing non-parametric tests. | After thirty patients have completed treatment.

SECONDARY OUTCOMES:
A qualitative evaluation will be scored as positive or negative. Twenty patients will allow this determination. | After twenty patients have recieved treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John D Davidson, MD, Principal Investigator — St. Luke's Hospital
Locations (2):
- United States (2):
  - St. Luke's Hospital, Chesterfield, Missouri
  - Mallinckrodt Institute of Radiology/Washington University Medical School, St Louis, Missouri